CLINICAL TRIAL: NCT00250328
Title: Evaluation of NiTi Laparoscopic Compression Anastomosis Clip (LapCAC) Device for Intra-Corporeal Lap-Colectomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO-CLP 52-01- HMO-CTIL
Record Dates: First submitted 2005-11-06; First posted 2005-11-08 (Estimated); Last update posted 2005-11-08 (Estimated); Status verified 2005-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

INTERVENTIONS:
Device: LapCAC Laparoscopic Compression Anastomosis Clip

SUMMARY:
The study involves adult subject requiring colonic anastomosis following laparoscopic intra-corporeal surgery. The anastomosis will be performed by using nitinilclip by the LapCAC device instead of staplers.

Endpoints: safety-Functioning secured anastomosis and no occurrence of adverse event related to device use.

The efficacy endpoint of this study includes clinical evaluation of characteristic parameters related to intestinal surgeries.

Discharge day (or ready-for-discharge) Proven anastomotic leak rate (clinically or radiological) Stenosis / stricture at anastomosis Patient recovery level will be assessed every day during hospitalization and in the follow up visits.

DETAILED DESCRIPTION:
The following steps are to be performed during the NiTi LapCAC surgical procedure.

1. Prophylactic antibiotic - as per specific department regimen.
2. Bowel preparation will be performed one-day prior to surgery. The preparation will included Sofodex solution combined with oral neomycin.
3. Aanticoagulation tratment prior surgery- as per specific department regimen.
4. Routine general anesthesia according to standard operation room procedure.
5. Prepare the surgery area according to routine procedure with soap and alcohol. Insert the trocars.
6. Align the two ends of bowel side-by-side in the same direction or in the opposite direction. Seal the ends with staples leaving blind loop of no less than 2.5 cm. (1 inch) and make two small enterotomies.
7. The Clip mounted on the Applier should be cooled by immersing it in ice-cold sterile saline bath for at least 20 seconds.
8. Place the open clip into the prepared enterotomies, each clip coil in one enterotomy.
9. Approximating body temperature, the coils will recover its programmed shape applying pressure on the tissue.
10. Closure (staple line and enterotomies): closure of the enterotomies with or without suture inversion of staple lines will be done by using Vicryl suture 3-0 or other absorbable suture. Postoperative care will be as for conventional treatment.
11. Post operative treatment will be according to the department regimen and in relation to the patient condition.

The following baseline variables will be recorded for all patients:

1. Demographics, including: gender, age, race, weight and height (BMI), ASA status.
2. Background of disease - presentation, and TNM stage, etc.
3. Region of excised colon.
4. Metastasis yes/no where.
5. Co-morbidities:

   Cardiac- (Ischemic heart disease (IHD), Congestive heart failure (CHF), NYHA Classification I,II,III,IV).

   Respiratory- Asthma, Obstructive pulmonary disease (OPD). Diabetes- Type 1(insulin-dependent diabetes), Type 2 (non-insulin-dependent diabetes).

   hepatic- Cirrhosis. Alcohol Smoking.
6. Medications.

Follow-up evaluation will be performed every day during hospitalization and one-month, three months and six months post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age over 18 years.
2. Patient schedule for colonic surgery which requires a bowel anastomosis (right colon, left colon, sigma).
3. Patient is able to understand and to sign the Informed Consent Form.

Exclusion Criteria:

1. Patient has known allergy to nickel.
2. Emergency procedure, i.e. patients with bowel obstruction, bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischaemic bowel, carcinomatosis.
3. Patients with Crohn's disease needed more than one anastomosis.
4. Patient underwent previous major abdominal surgery.
5. Patients under steroid treatment.
6. Patient albumin level less than 3 g/dl
7. Patients under immuno-suppression or cytotoxic treatment.
8. Patients who are participating in another trial which may affect the outcomes data on this study.
9. Patients with contraindications to general anaesthesia.
10. Patients who refuse consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-01

PRIMARY OUTCOMES:
Functioning anastomosis without leaks or obstructions

SECONDARY OUTCOMES:
Functioning anastomosis without stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Matter, MD, Principal Investigator — Benei-Zion Medical Center
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel